CLINICAL TRIAL: NCT04748328
Title: Comparison Effectiveness Analysis Between ACL Reconstruction and Rehabilitation in Peripheral and Main Capital of Indonesia
Brief Title: Comparison Effectiveness Analysis Between ACL Reconstruction and Rehabilitation in Peripheral and Main Capital in Indonesia
Acronym: Cetjap-Asin
Status: Active, not recruiting | Type: Observational
Sponsor: Universitas Riau (Other)
Responsible Party: Principal Investigator, Romy Deviandri, dr, Universitas Riau
Other Study IDs: KET-894
Record Dates: First submitted 2021-01-26; First posted 2021-02-10 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACL Reconstruction Group: This group received reconstruction treatment in Cipto Mangunkusumo Hospital, Gatot Subroto Hospital, Hasan Sadikin Hospital
  Interventions: Procedure: ACL Reconstruction surgery and Rehabilitation Treatment
- Rehabilitation Group: This group received rehabilitation treatment with optional delayed reconstruction if needed in Arifin Achmad Hospital, Pekanbaru
  Interventions: Procedure: ACL Reconstruction surgery and Rehabilitation Treatment

INTERVENTIONS:
Procedure: ACL Reconstruction surgery and Rehabilitation Treatment — ACL Reconstruction surgery is a procedure to treat ACL injury by replacing the torn ligament with another. ACL Rehabilitation treatment is a procedure to treat ACL injury by muscle strengthening and exercise

SUMMARY:
The study was a prospective observational analysis of cases with complete ACL tears. A study was conducted between February 2021 to December 2024. All the patients attending those hospitals' emergency or outpatient departments (OPD) with knee injuries were evaluated for an ACL tear. Patients who meet inclusion criteria and consent to participate in the study will be observed for two years. Patients in Arifin Achmad Hospital Pekanbaru will follow rehabilitation treatment and optional delayed reconstruction after 12 weeks if needed, while patients in some hospitals in Jakarta and Bandung (Cipto Mangunkusumo Hospital, Gatot Subroto Army Hospital, Hasan Sadikin Hospital) will perform early reconstruction treatment. After receiving informed consent, all subjects received a self-administered patient questionnaire containing the International Knee Documentation Committee (IKDC) score, EQ5D3L, and Tegner Activity Level (TAL) scores. These questionnaires will be measured at 0, 12, 24, 48, and 96 weeks. Clinical value of the Lachman test and pivot shift test will be performed. One independent orthopedic surgeon will keep all records and evaluate the results. All costs for the treatment will be accounted for.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 40 years
2. Either sex
3. Isolated ACL tear not more than six weeks old to a previously uninjured knee or less than six months with showing acute symptoms (inflammation, swelling, knee effusion)
4. Tegner Activitiy Level of 5-9.

Exclusion criteria

1. Professional athletes or military
2. Collateral ligament rupture
3. Full-thickness cartilage lesion visualized
4. TAL below 5
5. Meniscal tear grade III on MRI.
6. Pregnancy
7. A history of deep vein thrombosis (DVT) or a disorder of the coagulative system
8. Claustrophobia
9. General systemic disease affecting physical function, any other condition or treatment interfering with the completion of the trial, including patients with metal devices or motion disorders
10. Hyperlaxity with a Beighton score of more than 4

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Young active population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Questionnaire of International Knee Documentation Committee (IKDC Questionnaire) | IKDC questionnaire was measured at pre operation (0 month), 3rd month, 6th month, 12th month, 24th month
  IKDC is a subjective patient reported outcome measure for knee specific disease. Scoring in range 0-100, which 0 is lowest score, and 100 is a highest score

SECONDARY OUTCOMES:
Change of Lachman Test | at pre operation (0 month), 12th month, 24th month
  Lachman test was measured by passive movement of the knee at 30 degree of flexion, Grade 1: 3-5mm translation of the tibia Grade 2: 5-10 mm more translation of the tibia Grade 3: translation of the tibia more than 10mm
Change of Pivot shift test | at pre operation (0 month),12th month, 24th month
  Pivot shift test was measured by valgus and slowly flexion the knee, Grade 1: gentle twisting slide with tibia twisting internally maximally Grade 2: Clunk with tibia in neutral position Grade 3: painless glide for examiner and patient
Change of Questionnaire of EQ5D | at pre operation (0 month),12th month, 24th month
  The EQ5D questionnaire is a generic patient-reported outcome measure for measuring a patient's quality of life. Its scores range from -0,865 to 1 in the Indonesian population particularly.
Total cost of treatment | at 12th and 24 months
  Total cost for surgery treatment or rehabilitation treatment in Rupiah (Indonesian currency). Cost was taken account by direct interview to the patient and direct observation to medical account in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Arifin Achmad Hospital, Pekanbaru, Riau, Indonesia

IPD SHARING:
Plan to Share IPD: No